CLINICAL TRIAL: NCT03894332
Title: Electrical Impedance Tomography During Spontaneous Breathing Trial and Extubation Failure in Critically Ill Patients: an Observational Study
Brief Title: Lung Impedetiometric Modification in SBT and Extubation Failure
Acronym: CPAP2-EIT
Status: Completed | Type: Observational
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Federico Longhini, Associate Professor, University Magna Graecia
Other Study IDs: CPAP2EIT
Record Dates: First submitted 2019-02-10; First posted 2019-03-28 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Weaning Failure; Mechanical Ventilation Complication

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- SBT Success: Patients took part of this cohort when succeeding the Spontaneous Breathing Trial (SBT).
  Interventions: Diagnostic Test: Electrical Impedance Tomography (EIT)
- SBT Failure: Patients took part of this cohort when failing the Spontaneous Breathing Trial (SBT).
  SBT Failure is defined by one or more of the following criteria occurring during the SBT:
  1. loss of ≥ 2 points of Glasgow Coma Scale
  2. respiratory rate/ tidal volume ≥105 breaths/min/L
  3. arterial partial pressure of oxygen ≤60 mmHg on inspired oxygen fraction (FiO2) ≥0.5 and/or pH <7.32 or a decrease in pH ≥0.07 units at the end of the SBT
  4. systolic Blood Pressure <90 mmHg or ≥180 mmHg or increased by ≥20%
  5. Heart Rate >140 beats/min or increased by 20%
  6. onset of major heart arrhythmias, or electrocardiographic signs of cardiac ischemia
  7. Respiratory Rate ≥35 breaths/min or increased by ≥50%
  8. increased effort, respiratory distress (as indicated by diaphoresis, accessory respiratory muscles recruitment, facial signs of distress and/or paradoxical breath)
  Interventions: Diagnostic Test: Electrical Impedance Tomography (EIT)
- Extubation Success: Patients took part of this cohort when, after extubation, did not need continuous positive airways pressure (CPAP), non invasive ventilation (NIV) or reintubation within 48 hours.
  Interventions: Diagnostic Test: Electrical Impedance Tomography (EIT)
- Extubation Failure: Need for continuous positive airways pressure (CPAP), non invasive ventilation (NIV) or reintubation within 48 hours from extubation, as defined by:
  1. Respiratory Rate >25 breaths/min for 2 hours
  2. Heart Rate >140 beats/min or sustained increase or decrease >20%
  3. clinical signs of respiratory muscle failure
  4. arterial partial pressure of oxygen (PaO2) <80 mmHg on inspired oxygen fraction (FiO2) ≥50%
  5. Arterial partial pressure of carbon dioxide >45 mmHg with pH <7.33
  Interventions: Diagnostic Test: Electrical Impedance Tomography (EIT)

INTERVENTIONS:
Diagnostic Test: Electrical Impedance Tomography (EIT) — After enrollment, a silicon EIT belt of proper size with 16 electrodes was placed around the patient's chest between the 4th and 6th intercostal spaces, and connected to the EIT device. All patients were ventilated in Pressure Support Ventilation (PSV) mode, with a dedicated ventilator connected to the EIT device.
  We acquired 5-min EIT data records at baseline (during PSV), during the first (SBT_0) and the last (SBT_30) 5 minutes of SBT, and, when the patient was extubated, during spontaneous breathing soon after (SB_0) and 30 minutes after extubation (SB_30).
  EIT and ventilator data were recorded at a sample of 20 Hz. The last 3 minutes of each record were analyzed.
  We measured respiratory rate (RR); Vt changes from baseline, expressed as percent (dVt%); dEELI variations from baseline, expressed in mL; the Global Inhomogeneity index (GI); Impedance ratio (IR) and the Center of Ventilation (CoV).

SUMMARY:
Weaning is the entire process aimed at liberating patients from mechanical ventilation and endotracheal intubation. Weaning should be considered as early as possible in order to reduce the time spent in invasive mechanical ventilation (iMV), which is associated with morbidity and mortality. To verify if patients are ready to be extubated, a spontaneous breathing trial (SBT) is performed. At this stage some clinical indices and objective parameters are evaluated, such as the breathing pattern, gas exchange, haemodynamic stability and patient's comfort. In case of SBT success, the patient can be extubated. However, a post-extubation respiratory failure can occur within the first 48 hours after extubation, thus making extubation unsuccessful. Some patients considered at risk for post-extubation respiratory failure benefit from the application of non-invasive ventilation (NIV) after extubation. Early characterization of these patients is crucial to improve their clinical outcomes.

Electrical Impedance Tomography (EIT) has been introduced in clinical practice as a non-invasive bedside monitoring tool to evaluate the aeration and ventilation of different lung regions. EIT has been proposed to guide ventilator settings adjustments in critically ill patients and to monitor prolonged weaning. However, the potential of EIT to assess SBT and after extubation in a general ICU population has never been evaluated insofar.

The present study aims to describe the modifications of lung aeration, ventilation and inhomogeneity occurring during SBT and after extubation in a general population of critically ill patients at the first SBT attempt.

ELIGIBILITY:
Inclusion Criteria:

* Glasgow Coma Scale ≥8
* presence of clearly audible cough during suctioning with need for tracheal suctioning ≤2/hour
* normal sodium blood values
* core temperature <38.5° during the previous 8 hours
* Arterial partial pressure of oxygen to inspired oxygen fraction (PaO2/FiO2) ≥200 mmHg, with a Positive End Expiratory Pressure ≤5 cmH2O and FiO2 ≤0.4
* stable cardiovascular status (i.e., HR ≤140 beats/min, sBP between 90 and 160 mmHg without need for vasopressin, epinephrine or norepinephrine infusion, or with dopamine or dobutamine infusion ≤5 mcg/kg/min)
* cuff leak volume >110 mL

Exclusion Criteria:

* major heart arrhythmias or cardiac ischemia
* pneumothorax or emphysema
* recent (1 week) thoracic surgery
* presence of chest burns
* pregnancy
* inclusion in other research protocols

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We considered eligible any critically ill patient ≥18 years receiving invasive Mechanical Ventilation for at least 48 hours through an orotracheal tube, ready for the first Spontaneous Breathing Trial attempt, and met at least one criteria for increased risk of extubation failure.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-06-27 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Change of end-expiratory lung impedance (dEELI) from baseline at first 5 minute of Spontaneous Breathing Trial (SBT_0) | At 5 minutes of Spontaneous Breathing Trial (SBT)
  change from baseline, expressed in mL, of the end expiratory lung volume as assessed through electrical impedance tomography
Change of end-expiratory lung impedance (dEELI) from baseline at last 5 minute of Spontaneous Breathing Trial (SBT_30) | At the last 5 minutes of Spontaneous Breathing Trial (SBT)
  change from baseline, expressed in mL, of the end expiratory lung volume as assessed through electrical impedance tomography
Change of end-expiratory lung impedance (dEELI) from baseline at first 5 minute after extubation (SB_0) | At 5 minutes after extubation
  change from baseline, expressed in mL, of the end expiratory lung volume as assessed through electrical impedance tomography
Change of end-expiratory lung impedance (dEELI) from baseline at last 30 minute after extubation (SB_30) | At 30 minutes after extubation
  change from baseline, expressed in mL, of the end expiratory lung volume as assessed through electrical impedance tomography
Change of tidal volume in percentage (dVt%) from baseline at last 5 minute of SBT (SBT_0) | At 5 minutes of spontaneous breathing trial (SBT_0)
  change from baseline, expressed in percentage, of the end expiratory lung volume as assessed through electrical impedance tomography
Change of tidal volume in percentage (dVt%) from baseline from baseline at 30 minute of Spontaneous Breathing Trial (SBT_30) | At the last 5 minutes of Spontaneous Breathing Trial (SBT) (SBT_30)
  change from baseline, expressed in percentage, of the end expiratory lung volume as assessed through electrical impedance tomography
Change of tidal volume in percentage (dVt%) from baseline after 5 minutes from extubation (SB_0) | At 5 minutes after extubation (SB_0)
  change from baseline, expressed in percentage, of the end expiratory lung volume as assessed through electrical impedance tomography
Change of tidal volume in percentage (dVt%) from baseline at last 30 minute after extubation (SB_30) | At 30 minutes after extubation (SB_30)
  change from baseline, expressed in percentage, of the end expiratory lung volume as assessed through electrical impedance tomography
Inhomogeneity Index (GI) at baseline | At baseline during Pressure Support Ventilation
  Inhomogeneity Index (GI) as assessed through electrical impedance tomography
Inhomogeneity Index (GI) after 5 minutes of the Spontaneous Breathing Trials (SBT_0) | At 5 minutes of Spontaneous Breathing Trial (SBT_0)
  Inhomogeneity Index (GI) as assessed through electrical impedance tomography
Inhomogeneity Index (GI) after 30 minutes of the Spontaneous Breathing Trials (SBT_30) | At 30 minutes of Spontaneous Breathing Trial (SBT_30)
  Inhomogeneity Index (GI) as assessed through electrical impedance tomography
Inhomogeneity Index (GI) after 5 minutes from extubation (SB_0) | At 5 minutes after extubation (SB_0)
  Inhomogeneity Index (GI) as assessed through electrical impedance tomography
Inhomogeneity Index (GI) after 30 minutes from extubation (SB_30) | At 30 minutes after extubation (SB_30)
  Inhomogeneity Index (GI) as assessed through electrical impedance tomography

SECONDARY OUTCOMES:
Arterial Blood Gases at baseline | At baseline during Pressure Support Ventilation
  Arterial Blood was sampled for gas analysis
Arterial Blood Gases at SBT_30 | At 30 minutes of Spontaneous Breathing Trial (SBT_30)
  Arterial Blood was sampled for gas analysis
Arterial Blood Gases at SB_30 | At 30 minutes after extubation (SB_30)
  Arterial Blood was sampled for gas analysis
the ratio between respiratory rate (RR) and tidal volume (Vt) (RR/Vt) at baseline | At baseline during Pressure Support Ventilation
  the ratio between respiratory rate (RR) and tidal volume (Vt) (RR/Vt)
the ratio between respiratory rate (RR) and tidal volume (Vt) (RR/Vt) at 5 minutes of Spontaneous Breathing Trial (SBT_0) | At 5 minutes of Spontaneous Breathing Trial (SBT_0)
  the ratio between respiratory rate (RR) and tidal volume (Vt) (RR/Vt)
the ratio between respiratory rate (RR) and tidal volume (Vt) (RR/Vt) at SBT_30 | At 30 minutes of Spontaneous Breathing Trial (SBT_30)
  the ratio between respiratory rate (RR) and tidal volume (Vt) (RR/Vt)
the ratio between respiratory rate (RR) and tidal volume (Vt) (RR/Vt) at 5 minutes after extubation (SB_0) | At 5 minutes after extubation (SB_0)
  the ratio between respiratory rate (RR) and tidal volume (Vt) (RR/Vt)
the ratio between respiratory rate (RR) and tidal volume (Vt) (RR/Vt) at 30 minutes after extubation (SB_30) | At 30 minutes after extubation (SB_30)
  the ratio between respiratory rate (RR) and tidal volume (Vt) (RR/Vt)

CONTACTS AND LOCATIONS:
Overall Officials: Federico Longhini, Principal Investigator — Intensive Care Unit, University Hospital Mater Domini, Department of Medical and Surgical Sciences, Magna Graecia University

IPD SHARING:
Plan to Share IPD: Yes
The full protocol, datasets used and analysed during the current study are available on reasonable request at longhini.federico@gmail.com.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available from paper publication without any closing data

REFERENCES:
- [Background] Boles JM, Bion J, Connors A, Herridge M, Marsh B, Melot C, Pearl R, Silverman H, Stanchina M, Vieillard-Baron A, Welte T. Weaning from mechanical ventilation. Eur Respir J. 2007 May;29(5):1033-56. doi: 10.1183/09031936.00010206. PMID 17470624
- [Background] Nava S, Gregoretti C, Fanfulla F, Squadrone E, Grassi M, Carlucci A, Beltrame F, Navalesi P. Noninvasive ventilation to prevent respiratory failure after extubation in high-risk patients. Crit Care Med. 2005 Nov;33(11):2465-70. doi: 10.1097/01.ccm.0000186416.44752.72. PMID 16276167
- [Background] Ferrer M, Sellares J, Valencia M, Carrillo A, Gonzalez G, Badia JR, Nicolas JM, Torres A. Non-invasive ventilation after extubation in hypercapnic patients with chronic respiratory disorders: randomised controlled trial. Lancet. 2009 Sep 26;374(9695):1082-8. doi: 10.1016/S0140-6736(09)61038-2. Epub 2009 Aug 12. PMID 19682735
- [Background] Ferrer M, Valencia M, Nicolas JM, Bernadich O, Badia JR, Torres A. Early noninvasive ventilation averts extubation failure in patients at risk: a randomized trial. Am J Respir Crit Care Med. 2006 Jan 15;173(2):164-70. doi: 10.1164/rccm.200505-718OC. Epub 2005 Oct 13. PMID 16224108
- [Background] El-Solh AA, Aquilina A, Pineda L, Dhanvantri V, Grant B, Bouquin P. Noninvasive ventilation for prevention of post-extubation respiratory failure in obese patients. Eur Respir J. 2006 Sep;28(3):588-95. doi: 10.1183/09031936.06.00150705. Epub 2006 May 31. PMID 16737982
- [Background] Vianello A, Arcaro G, Braccioni F, Gallan F, Marchi MR, Chizio S, Zampieri D, Pegoraro E, Salvador V. Prevention of extubation failure in high-risk patients with neuromuscular disease. J Crit Care. 2011 Oct;26(5):517-524. doi: 10.1016/j.jcrc.2010.12.008. Epub 2011 Jan 26. PMID 21273033
- [Background] Ornico SR, Lobo SM, Sanches HS, Deberaldini M, Tofoli LT, Vidal AM, Schettino GP, Amato MB, Carvalho CR, Barbas CS. Noninvasive ventilation immediately after extubation improves weaning outcome after acute respiratory failure: a randomized controlled trial. Crit Care. 2013 Mar 4;17(2):R39. doi: 10.1186/cc12549. PMID 23497557
- [Background] Meade M, Guyatt G, Cook D, Griffith L, Sinuff T, Kergl C, Mancebo J, Esteban A, Epstein S. Predicting success in weaning from mechanical ventilation. Chest. 2001 Dec;120(6 Suppl):400S-24S. doi: 10.1378/chest.120.6_suppl.400s. PMID 11742961
- [Background] Costa EL, Lima RG, Amato MB. Electrical impedance tomography. Curr Opin Crit Care. 2009 Feb;15(1):18-24. doi: 10.1097/mcc.0b013e3283220e8c. PMID 19186406
- [Background] Frerichs I, Amato MB, van Kaam AH, Tingay DG, Zhao Z, Grychtol B, Bodenstein M, Gagnon H, Bohm SH, Teschner E, Stenqvist O, Mauri T, Torsani V, Camporota L, Schibler A, Wolf GK, Gommers D, Leonhardt S, Adler A; TREND study group. Chest electrical impedance tomography examination, data analysis, terminology, clinical use and recommendations: consensus statement of the TRanslational EIT developmeNt stuDy group. Thorax. 2017 Jan;72(1):83-93. doi: 10.1136/thoraxjnl-2016-208357. Epub 2016 Sep 5. PMID 27596161
- [Background] Zhao Z, Peng SY, Chang MY, Hsu YL, Frerichs I, Chang HT, Moller K. Spontaneous breathing trials after prolonged mechanical ventilation monitored by electrical impedance tomography: an observational study. Acta Anaesthesiol Scand. 2017 Oct;61(9):1166-1175. doi: 10.1111/aas.12959. Epub 2017 Aug 17. PMID 28832898
- [Background] Bickenbach J, Czaplik M, Polier M, Marx G, Marx N, Dreher M. Electrical impedance tomography for predicting failure of spontaneous breathing trials in patients with prolonged weaning. Crit Care. 2017 Jul 12;21(1):177. doi: 10.1186/s13054-017-1758-2. PMID 28697778
- [Background] Navalesi P, Frigerio P, Moretti MP, Sommariva M, Vesconi S, Baiardi P, Levati A. Rate of reintubation in mechanically ventilated neurosurgical and neurologic patients: evaluation of a systematic approach to weaning and extubation. Crit Care Med. 2008 Nov;36(11):2986-92. doi: 10.1097/CCM.0b013e31818b35f2. PMID 18824909
- [Background] Yang KL, Tobin MJ. A prospective study of indexes predicting the outcome of trials of weaning from mechanical ventilation. N Engl J Med. 1991 May 23;324(21):1445-50. doi: 10.1056/NEJM199105233242101. PMID 2023603
- [Background] Zhao Z, Moller K, Steinmann D, Frerichs I, Guttmann J. Evaluation of an electrical impedance tomography-based Global Inhomogeneity Index for pulmonary ventilation distribution. Intensive Care Med. 2009 Nov;35(11):1900-6. doi: 10.1007/s00134-009-1589-y. Epub 2009 Aug 4. PMID 19652949
- [Derived] Longhini F, Maugeri J, Andreoni C, Ronco C, Bruni A, Garofalo E, Pelaia C, Cavicchi C, Pintaudi S, Navalesi P. Electrical impedance tomography during spontaneous breathing trials and after extubation in critically ill patients at high risk for extubation failure: a multicenter observational study. Ann Intensive Care. 2019 Aug 13;9(1):88. doi: 10.1186/s13613-019-0565-0. PMID 31410738